

Title: AGRYLIN Capsules 0.5mg Drug Use Results Survey

NCT Number: NCT03625895

Statistical analysis plan Approve Date: 26-SEP-2019

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

Named persons or organizations associated with the study.

Patient identifiers within the text, tables, or figures or in by-patient data listings.

Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.

Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

### STATISTICAL ANALYSIS PLAN

| Protocol No.: | SHP422-406 |
|---|---|
| Protocol Title: | AGRYLIN Capsules 0.5mg Drug Use Results Survey |
| Drug: | AGRYLIN Capsules 0.5mg |
| Sponsor: | Shire Japan KK Tekko Building 21 F 1-8-1 Marunouchi, Chiyoda-ku |
| | 1-8-1 Marunouchi, Chiyoda-ku |
| | Tokyo 1000005 Japan |
| Version No. and Date | Version 3.0, Date 26SEP2019 |

| 77 ' 37 | D 'II' | A 41 ( ) | LCC . |
|---|---|---|---|
| Version No: | Document History Description of Undate | Author(s) | Effective |
| | Description of Update | | Date |
| 1.0 | N/A | PPD | 13AUG2015 |
| | Se | | |
| 2.0 | Add new subject population sets. | PPD | 11JAN2018 |
| | Add Final Analysis Efficacy. | | |
| | Add important items for investigation. | | |
| 3.0 | Updated MedDRA version. | PPD | 26SEP2019 |
| | Updated SAS version. | | |
| Property of Lakeda. F | SK . | | |
| 8 to 6 | | | |

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 1 of 29



### **TABLE OF CONTENTS**

| TAB | BLE OF CONTENTS | 2 |
|---|---|---|
| LIST | OF TABLES | 4 |
| ABB | BREVIATIONS | 5 |
| 1. | INTRODUCTION | 6 |
| 2. | SURVEY DESIGN General Survey Design Randomization Blinding | 7 |
| 2.1 | General Survey Design | <b>?</b> 7 |
| 2.2 | Randomization | 7 |
| 2.3 | Blinding | 7 |
| 2.4 | Schedule of Assessments Determination of Sample Size Multiplicity Adjustments for Type I Error Control | 8 |
| 2.5 | Determination of Sample Size | 9 |
| 2.6 | Multiplicity Adjustments for Type I Error Control | 9 |
| 3. | OBJECTIVES | 10 |
| 4. | SUBJECT POPULATION SETS | 11 |
| 4.1 | Enrolled Sets. | 11 |
| ۷ | 4.1.1 The Pre-Data Lock Point Enrolled Set | 11 |
| ۷ | 4.1.2 The Overall Enrolled Set | 11 |
| 4.2 | 4.1.2 The Overall Enrolled Set | 11 |
| ۷ | 4.2.1 The Pre-Data Lock Point Safety Analysis Set | |
| ۷ | 4.2.2 The Overall Safety Analysis Set | |
| 4.3 | Efficacy Analysis Sets | |
| ۷ | 4.3.1 The Pre-Data Dock Point Efficacy Analysis Set | 11 |
| 2 | 4.3.2 The Overall Efficacy Analysis Set | |
| 5. | SUBJECT DISPOSITION | 12 |
| 6. | PROTOCOL DEVIATIONS | 13 |
| 7. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 14 |
| 8.01 | EXTENT OF EXPOSURE | 15 |
| 8.1 | Exposure to Agrylin | 15 |
| 9. | CONCOMITANT MEDICATION | 16 |
| 10. | EFFICACY ANALYSES | 17 |

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02, Effective Date: 26 Sep 2019

Page No.: 2 of 29



| 10.1 | Primary Efficacy Endpoint(s) and Analysis | 17 |
|---|---|---|
| 10.2 | Exploratory Efficacy Endpoint(s) and Analyses | |
| 10.3 | For Final Analysis Efficacy Endpoint(s) and Analyses | 17 |
| 11. | SAFETY ANALYSES | 19 |
| 11.1 | Adverse Events | 19 |
| 11.2 | Clinical Laboratory Variables | ( |
| 11.3 | Vital Signs | 4 1 |
| 11.4 | | |
| 11.5 | Electrocardiogram Other Safety Variables | 20 |
| 12. | ADVERSE EVENTS OF SPECIAL INTEREST (IMPORTANT ITEMS FOR | |
| 13. | INVESTIGATION) | 22 |
| 14. | DATA MONITORING/REVIEW COMMITTEE | 23 |
| 15. | DATA MONITORING/REVIEW COMMITTEE COMPUTER METHODS CHANGES TO ANALYSES SPECIFIED IN PROTOCOL | 24 |
| 16. | CHANGES TO ANALTSES STEER IED INTROTOCOL | 23 |
| 17. | DATA HANDLING CONVENTIONS | 26 |
| 17.1 | General Data Reporting Conventions | 26 |
| 17.2 | Derived Efficacy Endpoints | 26 |
| 17.3 | Repeated or Unscheduled Assessments of Efficacy and Safety Parameters | 26 |
| 17.4 | Missing Date of Agrylin | 26 |
| 17.5 | Missing Date Information for Concomitant Medications | 26 |
| | .5.1 Incomplete Start Date | |
| 17 | .5.2 Incomplete Stop Date | 27 |
| 17.6 | Missing Date Information for Adverse Events | 28 |
| 17 | .6.1 Incomplete Start Date | 28 |
| 17 | .6.2 Incomplete Stop Date | 28 |
| 17.7 | Missing Severity Assessment for Adverse Events | 28 |
| 17.80 | Missing Relationship to Agrylin for Adverse Events | 28 |
| 17.9 | Character Values of Clinical Laboratory Variables | 28 |
| 17.10 | Baseline Values | 28 |
| 18. | REFERENCES | 29 |

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02, Effective Date: 26 Sep 2019

Page No.: 3 of 29



### LIST OF TABLES

| LIST OF TABLES | |
|---|---|
| Table 1: Schedule of Assessments | |
| Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02. Ffective Date: 26 Sep 2019 Page No.: 4 of 292 | 500 |
| Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02, Effective Date: 26 Sep 2019 Page No.: 4 of 29 | |



### **ABBREVIATIONS**

arombocythemia
acerstitial lung disease
Medical Dictionary for Regulatory Activities
Pharmaceuticals and Medical Devices Agency
preferred term
statistical analysis plan
standard deviation
system organ class
treatment-emergent adverse event AΕ **BMI CRF** CI

**DURS** 

**ECG** ЕСНО

ET ILD

MedDRA

**PMDA** 

PT

SAP SD Property of Takeda. For non-commercial use of Property of Takeda. SOC

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 5 of 29



#### 1. INTRODUCTION

properly of Takeda. For non-commercial use only and subject to the applicable of the property of takeda.

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 6 of 29



#### 2. SURVEY DESIGN

#### 2.1 **General Survey Design**

FINS OF USE This is a Drug Use Results Survey (DURS) of Agrylin (anagrelide hydrochloride) in the postmarketing phase in patients diagnosed with Essential Thrombocythemia (ET).

Planned implementation period of this survey is as follows:

- 1. Implementation period: from product approval until the approval condition regarding implementation of the all case survey is removed. 1
- 2. Patient registration: from the approval to the approval condition regarding to all case survey is removed. However, for all patients who were prescribed Agrylin prior to 31 May, 2015, all CRFs must be completed and included in the analysis. Patients who were ay, 2
  2 or 31 M
  proval cond

  Lecived treatment with Agryl
  ar.

  .ndomization
  .ticable to this survey.

  Blinding

  Not applicable to this survey.

  Adv. 2
  2 or 31 M
  proval cond

  Lecived treatment with Agryl
  ar.

  .ndomization
  .ticable to this survey.

  Blinding

  Not applicable to this survey.

  Property 4 decived treatment with Agryl
  ar. prescribed Agrylin after 31 May, 2015, should be included in the analysis if CRF has already been completed. After 31 May, 2015, it is planned that only patient registration will continue until the approval condition is removed. All CRFs will be collected and

All patients who received treatment with Agrylin will be included in this survey and will be

<sup>1</sup> The implementation period is from the launch of XAGRID in Japan to receipt of approval from the Pharmaceuticals and Medical Devices Agency (PMDA) to discontinue the survey. At least 474 subjects must be registered and followed for 1-

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02, Effective Date: 26 Sep 2019

Page No.: 7 of 29



#### 2.4 **Schedule of Assessments**

Safety and efficacy data that are available as part of routine clinical practice related to the treatment with Agrylin will be investigated.

Table 1: **Schedule of Assessments** 

| | Danis de di | | Book 1 | | Во | ok 2 |
|---|---|---|---|---|---|---|
| | Registration<br>Form | Registration | Additional<br>Visit | 6 Month<br>visit | Additional<br>Visit | 12 Month<br>visit |
| Patient identification number | • | • | | | 76 | ) |
| Patient initials | • | | | | 70. | |
| Date of birth (Age) | • | • | | | 1100 | |
| Sex | • | • | | | 0// | |
| Race | | • | | a' | 2 | |
| Diagnosis of ET | | • | | 0, | | |
| JAK2 status | | • | | KILO | | |
| Testing for pathogenetic mutations | | • | ١ | | | |
| Bone marrow biopsies | | • | X | | | |
| Testing to rule out other hematological | | • | | | | |
| malignancies | | | | | | |
| Prior treatments for ET | | • 6 | 200 | | | |
| Medical history/Complication | | • > 9 | | | | |
| Echocardiogram (If Applicable) | | | • | • | • | • |
| Electrocardiogram (If Applicable) | | . 76 | • | • | • | • |
| Vital signs (Blood Pressure, Pulse) | | 77 • | • | • | • | • |
| Height | | • | | | | |
| Weight | 01 | • | • | • | • | • |
| Pregnancy status (Urinalysis) | 1,5 | • | • | • | • | • |
| Administration status | | • | • | • | • | • |
| Concomitant therapy | CO. | • | • | • | • | • |
| Safety (Adverse Event) | 30 | • | • | • | • | • |
| Efficacy (Platelet count) | Ψ | • | • | • | • | • |
| Date of Discontinuation/Reason for | · | | • | • | • | • |
| Discontinuation Discontinuation | | | | | | |
| Important Items for investigation | | • | • | • | • | • |
| (Cardiac disorders, QT/QTc | | | | | | |
| prolongation, Thrombohaemorrhage | | | | | | |
| events, Interstitial lung disease) | | | | | | |
| ET=essential thrombocytemia; JAK=Jan | nus-Activated Kinas | se; QTc=correcte | d QT interval | | | |
| Title: Statistical Analysis Plan Te | | ıt No.: RD FOI | RM-0111 | | S | hire |

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 8 of 29



#### 2.5 **Determination of Sample Size**

### **Target Patient Population**

All cases who received treatment with Agrylin.

### Target number of cases: 474 cases

150 USE It is estimated that 474 patients will be prescribed Agrylin at the end of the second year of marketing in Japan. This number suffices to potentially observe with 95% confidence interval entry and subject to the administrative of Lakeda. For noncommercial use only and subject to the appropriate of Lakeda. (CI) (exact binomial CI estimated by Clopper & Pearson method) common adverse events that are classified as important investigation items in this all-case survey; less common events such as interstitial lung disease (ILD) or some cardiac disorders (e.g., Torsade de

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02, Effective Date: 26 Sep 2019

Page No.: 9 of 29



#### 3. **OBJECTIVES**

Properly of Takeda. For non-commercial use only and subject to the applicable Terms of use

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 10 of 29



### 4. SUBJECT POPULATION SETS

The following populations are defined:

### 4.1 Enrolled Sets

The following two types of Enrolled Set are created.

### 4.1.1 The Pre-Data Lock Point Enrolled Set

The Pre-Data Lock Point (DLP) Enrolled Set will consist of all subjects in the Overall Enrolled Set who started treatment with Agrylin before May 31, 2015.

### 4.1.2 The Overall Enrolled Set

The Overall Enrolled Set will consist of all subjects who are enrolled in this survey.

### 4.2 Safety Analysis Sets

### 4.2.1 The Pre-Data Lock Point Safety Analysis Set

The Pre-DLP Safety Analysis Set will consist of all subjects in the Pre-DLP Enrolled Set (Section 4.1.1) who started treatment with Agrylin before May 31, 2015 and have provided any post-registration data.

# 4.2.2 The Overall Safety Analysis Set

The Overall Safety Analysis Set will consist of all subjects in the Overall Enrolled Set (Section 4.1.2) who have received at least one dose of Agrylin and have provided any post-registration data.

### 4.3 Efficacy Analysis Sets

### 4.3.1 The Pre-Data Lock Point Efficacy Analysis Set

The Pre-DLP Efficacy Analysis Set will consist of all subjects in the Pre-DLP Safety Analysis Set (Section 4.2.1) who started treatment with Agrylin before May 31, 2015 and have at least one post-baseline platelet count assessment.

### 4.3.2 The Overall Efficacy Analysis Set

The Overall Efficacy Analysis Set will consist of all subjects in the Overall Safety Analysis Set (Section 4.2.2) who have at least one post-baseline platelet count assessment.

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 11 of 29



Rev. 02, Effective Date: 26 Sep 2019

Page No.: 12 of 29



#### **6.** PROTOCOL DEVIATIONS

Prodety of Lakeda: For non-commercial use only and subject to the applicable Lennes of use Rev. 02, Effective Date: 26 Sep 2019

Page No.: 13 of 29



#### 7. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Continuous variables such as age, weight, and height will be summarized using the number of observations, mean, standard deviation (SD), median, minimum, and maximum values. Categorical variables such as age category and sex will be summarized using the number of observations and percentages.

Descriptive summaries of demographic and baseline characteristics will be presented for the Pre-DLP Safety Analysis Set (Section 4.2.1) and Overall Safety Analysis Set (Section 4.2.2).

The following demographic characteristics will be summarized in the tables: sex, age (years), age category and time since ET diagnosis (years) (calculated by [start date of Agrylin administration - date of ET diagnosis]/365.25).

In addition, the following baseline characteristics will be summarized in the tables: JAK-2 status (positive, negative, not done), prior thrombocythaemia therapy (no, yes, with subcategories anti-platelet therapy, ant-coagulant therapy, thrombolytic agent, and response [refractory/intolerant/other] for each subcategories and overall), weight (kg), height (m), body mass index (BMI, calculated by weight(kg) / height(m)^2), BMI category, platelet counts, platelet counts category, and pregnancy test result (positive, negative, not applicable) at baseline (registration visit).

Medical histories and complications will be coded using the Medical Dictionary for Regulatory Activities (MedDRA Ver22.0) and will be summarized by the following CRFspecified categories:

- Hepatic impairment (no, yes, missing, with categories of severity)
- Renal impairment (no, yes, missing, with categories of severity)
- Cardiac disorders (no, yes, missing)
- QT/QTc prolongation (no, yes, missing)
- Thrombohemorrhagic events (no, yes, missing)
- Interstitial lung disease (no, yes, missing)
- Others (no, yes, missing)

Property of Taken All demographic and other baseline characteristics will be listed.

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 14 of 29



#### 8. EXTENT OF EXPOSURE

#### 8.1 **Exposure to Agrylin**

Exposure to Agrylin will be summarized for the Pre-DLP Safety Analysis Set (Section 4.2.1) and Overall Safety Analysis Set (Section 4.2.2) in terms of following parameters. Descriptive statistics (n, mean, SD, minimum, median, and maximum) will be presented.

- Duration of exposure (days): the stop date of Agrylin administration the start date of Agrylin administration +1.
- Total dose (g): summation (over the different intervals of total daily doses) of ([stop date of Agrylin administration - start date of Agrylin administration + 1] x total daily dose (mg))/1000
- Average daily dose (mg/day): total dose (g) / duration of exposure (days) x 1000.

Subjects in the Overall and Pre-DLP Safety Analysis Sets whose total daily dose of Agrylin Property of Takeda. For non-commercial use only and suppose of takeda. exceeded 7mg/day will be similarly summarized.

The number and percentage of subjects who met each of these criteria will also be displayed.

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02, Effective Date: 26 Sep 2019

Page No.: 15 of 29



#### 9. CONCOMITANT MEDICATION

Concomitant medication is defined as any medication with a start date prior to the start date of Agrylin administration and continuing after the start date of Agrylin administration or with a start date between the dates of the start date and the stop date of Agrylin administration, inclusive. Any medication with the end date before the start date of Agrylin administration or the start date after the stop date of Agrylin administration will not be considered a concomitant medication.

Additional details related to missing or incomplete dates are addressed in Section 17.

Concomitant medication usage for the Pre-DLP Safety Analysis Set (Section 4.2.1) and Overall and Safety Analysis Set (Section 4.2.2) will be summarized by the number and proportion of subjects receiving each medication within each type of medication (anti-platelet erie my once. Takeda. For noncommercial use only and subject to therapies, anti-coagulant, thrombolytic agents, others) and generic name. Multiple medication usage by a subject in the same category will be counted only once.

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 16 of 29



### 10. EFFICACY ANALYSES

All efficacy analyses will be based on the Pre-DLP Efficacy Analysis Set (Section 4.3.1) and Overall Efficacy Analysis Set (Section 4.3.2). Baseline for all efficacy analyses is defined as the value for the efficacy assessment at the registration visit. Platelet count is the only efficacy parameter.

Descriptive statistics, consisting of the number of observations, the mean, the standard deviation, the median, and the minimum, and maximum values, will be presented, but no statistical tests will be performed.

### 10.1 Primary Efficacy Endpoint(s) and Analysis

The primary efficacy variable is platelet count, for which the absolute value will be summarized, by visit (Baseline, 1 Months, 3 Months, 6 Months, 9 Months, 12 Months), using descriptive statistics for the Efficacy Analysis Set.

### 10.2 Exploratory Efficacy Endpoint(s) and Analyses

Platelet counts will be similarly summarized for the Overall and Pre-DLP Efficacy Analysis Sets by age group ( $\leq$  17 [pediatric], 18-64,  $\geq$  65 [elderly]), baseline hepatic impairment group (yes, no, missing), baseline renal impairment group (yes, no, missing), baseline urine pregnancy test group (positive, negative), and by prior thrombocythemia therapy group (yes, no).

### 10.3 For Final Analysis Efficacy Endpoint(s) and Analyses

The control rate of platelet count will be summarized using the number of observations and percentages. The control rate of the platelet count is determined as follows.

| Baseline | Survey data after 91 days (3 months) after Agrylin administration | The control rate of the platelet count (600,000 / uL) |
|---|---|---|
| 600,000 / uL or more | less than 600,000 / uL | Achieved |
| 600,000 / uL or more | 600,000 / uL or more | Not achieved |
| less than 600,000 / uL | less than 600,000 / uL | Undecidable |
| less than 600,000 / uL | 600,000 / uL or more | Undecidable |

| Baseline | Survey data after 91 days (3 months) after Agrylin administration | The control rate of the platelet count (400,000 / uL) |
|---|---|---|
| 400,000 / uL or more | less than 400,000 / uL | Achieved |
| 400,000 / uL or more | 400,000 / uL or more | Not achieved |

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 17 of 29



| less than 400,000 / uL | less than 400,000 / uL | Undecidable |
|------------------------|------------------------|-------------|
| less than 400,000 / uL | 400,000 / uL or more | Undecidable |

| Rate of change | The control rate of the platelet count |
|---|---|
| (After Agrylin administration - Baseline) /Baseline * 100 | (50% decrease) |
| -50% or less | Achieved |
| more than -50% | Not achieved |
| Title: Statistical Analysis Plan Template, Document No.: Rev. 02. Effective Date: 26 Sep 2019 Page No.: 18 Sor 29 | RD FORM-0111 |
| Rev. 02, Effective Date: 26 Sep 2019 Page No.: 18 of 29 | S Control of the second of the |



#### 11. SAFETY ANALYSES

The safety analysis will be performed using the Pre-DLP Safety Analysis Set (Section 4.2.1) Terms of Use and Overall Safety Analysis Set (Section 4.2.2). Safety parameters include adverse events (AEs), vital signs, and electrocardiogram (ECG) parameters. For each safety parameter, the registration visit value will be used as the baseline value.

#### 11.1 **Adverse Events**

Adverse events will be coded using the MedDRA (appropriate version).

An AE (classified by PT) that occurs during the observation period will be considered a treatment-emergent adverse event (TEAE) if it has a start date on or after the start date of Agrylin administration or if it has a start date before the start date of Agrylin administration, but increases in severity on or after the start date of Agrylin administration. If more than 1 AE with the same PT is reported before the start date of Agrylin administration, then the AE with the greatest severity will be used as the benchmark for comparison to the AEs occurring during observation period under the PT. If a TEAE is determined to be related to Agrylin, it is classified as an Adverse Drug Reaction (ADR).

An overall summary of the number of subjects with TEAEs will be presented, including the number and percentage of subjects with any TEAEs, serious TEAEs, TEAEs related to Agrylin, TEAEs leading to dose interruption and TEAEs leading to drug withdrawal. The number and percentage of subjects reporting TEAEs will be tabulated by system organ class (SOC) and PT; by SOC, PT, and maximum severity. TEAEs considered related to Agrylin (ADRs) and serious TEAEs will also be summarized by SOC and PT. If more than 1 AE occurs with the same PT for the same subject, then the subject will be counted only once for that PT using the most severe and most related occurrence for the summarization by severity and by relationship with Agrylin

The number of subjects in the Overall and Pre-DLP Safety Analysis Sets with any TEAEs will also be summarized by Outcome.

• Age category (<= 17 [pediatric], 18 – 64, >= 65 [elderly])

(<= 17, 18 - 44, 45 - 54, 55 - 64, 65 - 74

• Baseline Hepatic impairment (\*\*\*
• Baseline P The number and percentage of subjects in the Overall and Pre-DLP Safety Analysis Sets with any TEAEs will also be summarized by the following background or baseline factors:

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 19 of 29



- Prior thrombocythaemia therapy (yes, no, missing)
- Other factors judged necessary (Details are described in TLF Shells)

Terms of Use In addition, the number and percentage of subjects reporting TEAEs will be tabulated by PT for each of the background or baseline factors listed below.

- Children (Aged Under 18 Years), Elderly (Aged 65 or Older)
- Pregnant
- Important Items for investigation (Hepatic Impairment, Renal desorder, Cardiac Disorders, QT/QTc Prolongation, Hematological Toxicity, Thrombohemorrhagic Events, Interstitial Lung Disease, Headache)

TEAEs with an incidence 1.00% or more are defined as "Major TEAEs" "Major TEAEs" will be tabulated by PT.

#### 11.2 **Clinical Laboratory Variables**

Except for platelet counts, laboratory tests are not mandatory for this survey and related data will be collected as available for the parameters relevant to AEs.

Laboratory test data will be listed only.

### 11.3 Vital Signs

Descriptive statistics for vital signs (e.g., systolic and diastolic blood pressure, pulse rate, and body weight) and their changes from baseline at each post-baseline visit (6 and 12 months visit) will be presented.

### 11.4 Electrocardiogram

Electrocardiogram is not mandatory test for this survey.

Electrocardiogram will be listed only if performed.

# Other Safety Variables

# **Echocardiogram (ECHO):**

An ECHO is not mandatory in this survey.

ECHO data will be listed only if performed.

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 20 of 29



### 12. ADVERSE EVENTS OF SPECIAL INTEREST (IMPORTANT **ITEMS FOR INVESTIGATION)**

applicable Terms of Use The following CRF-specified categories of AEs are termed "important items for investigation" for this survey.

- Cardiac disorder
- QT/corrected QT interval (QTc) prolongation
- Thrombohemorrhagic events
- Interstitial lung disease
- Haematological toxicity
- Headache

These important items for investigation will be summarized using the number and proportion of subjects together with the 2-sided 95% CIs (exact binomial CI estimated by Clopper & Pearson method) per post-treatment visit (6 Months, 12 Months) and overall for the Pre-DLP Safety Analysis Set (Section 4.2.1) and Overall Safety Analysis Set (Section 4.2.2).

ety .ing TEAl and reading and .For non-commercial use only and .Por non-commercial use of .Por non-commercial use .Por non-commer The number and percentage of subjects reporting TEAEs within each of these important items

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02, Effective Date: 26 Sep 2019

Page No.: 21 of 29



#### **13. INTERIM ANALYSIS**

Proofeth of Takeda: For non-commercial use only and subject to the applicable Terms of use

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 22 of 29



#### 14. DATA MONITORING/REVIEW COMMITTEE

Probeth of Lakeda: For non-commercial use only and subject to the applicable Lennes of use Rev. 02, Effective Date: 26 Sep 2019

Page No.: 23 of 29



#### 15. **COMPUTER METHODS**

properly of Takeda: For noncommercial use only and subject to the applicable Terms of use

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 24 of 29



### **16.** CHANGES TO ANALYSES SPECIFIED IN PROTOCOL

Prodety of Lakeda: For non-commercial use only and subject to the applicable Lennes of use Rev. 02, Effective Date: 26 Sep 2019

Page No.: 25 of 29



### 17. DATA HANDLING CONVENTIONS

### 17.1 General Data Reporting Conventions

Continuous variables will be summarized using the following descriptive statistics: n, mean, median, SD, minimum, maximum. Categorical and count variables will be summarized by the number of subjects (n) and the percent of subjects in each category. Percentages will be presented as whole numbers.

Refer to TFLs4Shire for rules on the number of decimal places to present data and p-values.

### 17.2 Derived Efficacy Endpoints

Not applicable for this survey.

# 17.3 Repeated or Unscheduled Assessments of Efficacy and Safety Parameters

The last observation within each reporting period (baseline, 6 month, 12 month) will be summarized. All assessments, including unscheduled, will be presented in the data listings.

### 17.4 Missing Date of Agrylin

Not applicable for this survey.

### 17.5 Missing Date Information for Concomitant Medications

For concomitant medication summaries, incomplete (i.e., partially missing) start date and/or stop date will be imputed. When the start date and the stop date are both incomplete for a subject, impute the start date first.

## 17.5.1 Incomplete Start Date

The following rules will be applied to impute the missing numerical fields. If the stop date is complete and the imputed start date is after the stop date, then the start date will be imputed using the stop date.

### Missing day and month

- If the year of the incomplete start date is the same as the year of the start date of Agrylin administration, then the day and month of the start date of Agrylin administration will be assigned to the missing fields
- If the year of the incomplete start date is before the year of the start date of Agrylin administration, then December 31 will be assigned to the missing fields
- If the year of the incomplete start date is after the year of the start date of Agrylin administration, then 01 January will be assigned to the missing fields.

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111 Rev. 02, Effective Date: 26 Sep 2019

Page No.: 26 of 29



### Missing month only

• The day will be treated as missing and both month and day will be replaced according to the above procedure.

### Missing day only

- If the month and year of the incomplete start date are the same as the month and year of the start date of Agrylin administration, then the day of the start date of Agrylin administration will be assigned to the missing day
- If either the year is before the year of the start date of Agrylin administration or if both years are the same but the month is before the month of the start date of Agrylin administration, then the last day of the month will be assigned to the missing day
- If either the year is after the year of the start date of Agrylin administration or if both years are the same but the month is after the month of the start date of Agrylin administration, then the first day of the month will be assigned to the missing day.

### 17.5.2 Incomplete Stop Date

The following rules will be applied to impute the missing numerical fields. If the imputed stop date is before the start date (imputed or non-imputed start date), then the imputed stop date will be equal to the start date.

### Missing day and month

- If the year of the incomplete stop date is the same as the year as of the stop date of Agrylin administration, then the day and month of the date of the stop date of Agrylin administration will be assigned to the missing fields
- If the year of the incomplete stop date is before the year of the stop date of Agrylin administration, then 31 December will be assigned to the missing fields
- If the year of the incomplete stop date is after the year of the stop date of Agrylin administration, then 01 January will be assigned to the missing fields.

### Missing month only

• The day will be treated as missing and both month and day will be replaced according to the above procedure.

# Missing day only

• If the month and year of the incomplete stop date are the same as the month and year of the stop date of Agrylin administration, then the day of the stop date of Agrylin administration will be assigned to the missing day

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 27 of 29



- If either the year is before the year of the stop date of Agrylin administration or if both years are the same but the month is before the month of the stop date of Agrylin administration, then the last day of the month will be assigned to the missing day
- an of Use If either the year is after the year of the stop date of Agrylin administration or if both years are the same but the month is after the month of the stop date of Agrylin administration, then the first day of the month will be assigned to the missing day.

#### 17.6 Missing Date Information for Adverse Events

For AEs, only incomplete (i.e., partially missing) start dates will be imputed.

### 17.6.1 **Incomplete Start Date**

The same rules as those provided in Section 17.5.1 will be followed.

#### 17.6.2 **Incomplete Stop Date**

If required per the protocol, the same rules as those provided in Section 17.5.2 will be followed.

#### 17.7 Missing Severity Assessment for Adverse Events

If severity is missing for an AE starting prior to the start date of Agrylin administration, then a severity of "Mild" will be assigned. If the severity is missing for an AE starting on or after the start date of Agrylin administration, then a severity of "Severe" will be assigned. The imputed values for severity assessment will be used for incidence summaries, while the actual values will be used in data listings.

### Missing Relationship to Agrylin for Adverse Events 17.8

If the relationship to Agrylin is missing for an AE starting on or after the start date of Agrylin administration, a causality of "Related" will be assigned. The imputed values for relationship to Agrylin will be used for incidence summaries, while the actual values will be presented in data listings.

#### 17.9 **Character Values of Clinical Laboratory Variables**

Not applicable for this survey.

### **Baseline Values** 17.10

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered pre-baseline, except for Adverse Events (AEs) and medications commencing on the reference start date, which will be considered post-baseline

Title: Statistical Analysis Plan Template, Document No.: RD FORM-0111

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 28 of 29



#### **REFERENCES 18.**

Probeth of Takeda: For non-commercial life only and subject to the applicable Terms of tiese

Rev. 02, Effective Date: 26 Sep 2019

Page No.: 29 of 29

